CLINICAL TRIAL: NCT04313257
Title: Monocular Action Video Game Versus Passive Occlusion In The Treatment Of Amblyopia: A Randomized Controlled Trial
Brief Title: Monocular Action Video Game Treatment of Amblyopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Politècnica de Catalunya (Other)
Collaborators: Hospital Mutua de Terrassa (Other); Parc Sanitari Sant Joan de Déu (Other)
Responsible Party: Principal Investigator, Laura Asensio Jurado, Principal Investigator, Universitat Politècnica de Catalunya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PhDLAJE1
Record Dates: First submitted 2020-03-08; First posted 2020-03-18 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Amblyopia; Amblyopia Occlusion; Unilateral Amblyopia; Anisometropic Amblyopia; Strabismic Amblyopia
Keywords: Action Video Games; Amblyopia treatment
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive Occlusion (Active Comparator): This arm will include those participants who will follow a daily occlusive treatment of 2 hours.
  Interventions: Other: Monocular Passive Occlusion
- Active Occlusion (Experimental): This arm will include patients who will be treated with monocular therapy with video-games of one hour on a daily regimen.
  Interventions: Other: Monocular Active Occlusion

INTERVENTIONS:
Other: Monocular Active Occlusion — Occlusion treatment of one hour daily with action video game.
  Arms: Active Occlusion
Other: Monocular Passive Occlusion — Occlusion treatment of two hour daily.
  Arms: Passive Occlusion

SUMMARY:
This study evaluates the effectiveness of the monocular treatment with action video-games in comparison with the occlusion therapy alone in amblyopic patients, and the satisfaction with the different evaluated treatments.

DETAILED DESCRIPTION:
Amblyopia is the condition in which there is a decrease in monocular visual acuity or, less frequently, binocular, in absence of structural anomalies or ocular pathology. It is a reversible condition that affects up to 5% of the population, and that is the result of an abnormal visual experience during the most sensitive period of visual development.

The aim of this study is reviewing, analyzing and, if applicable, updating the current treatment model for amblyopia.

A randomized clinical trial will be performed to evaluate the effectiveness of the monocular treatment with action video-games in comparison with the occlusion therapy alone in amblyopic patients, and the satisfaction with the different evaluated treatments. The participants will be distributed in two groups. The first group will include those participants who will follow a daily occlusive treatment and the second group will include patients who will be treated with monocular therapy with video-games.The sample will include subjects between 4 to 10 years old with a diagnosis of refractive and / or strabismic amblyopia.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-10 years old
* Anisometropic amblyopia
* Strabismic amblyopia or mixed
* Interocular visual acuity (VA) difference of at least 0.2 logMAR
* No history of eye surgery

Exclusion Criteria:

* Non-comitant and/or large constant strabismus (>30 prism diopters)
* Any ocular pathological condition or nystagmus

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline visual acuity (VA) at 14 hours , 28 hours , and 42 hours comparing passive occlusion vs active occlusion (with action video games). | Baseline and 14, 28 and 42 hours post treatment.
  Visual Acuity (VA in logMAR) will be evaluated by E Snellen Test through an Ipad and the app AmblyopiaVA. The AmblyopiaVA test is designed based on the standard protocol for measuring Visual Acuity in children with Amblyopia.The measure will be performed at 2 m.
Change from baseline stereopsis (ST) at 14 hours , 28 hours , and 42 hours comparing passive occlusion vs active occlusion (with action video games). | Baseline and 14, 28 and 42 hours post treatment.
  Stereopsis (ST in logMAR) will be evaluated by a Multiple Random Points test through an Ipad, the app StereoTAB and anaglyphic glasses. The measures will be performed at 50 cm.
Change from baseline contrast sensitivity function (CSF) at 14 hours , 28 hours , and 42 hours comparing passive occlusion vs active occlusion (with action video games). | Baseline and 14, 28 and 42 hours post treatment.
  The effect of treatment on Contrast Sensitivity Function (CSF in logMAR) will be evaluated by ClinicCFS test using sine grids of four different spatial frequencies: 3, 6, 12 and 18 cpd.

SECONDARY OUTCOMES:
Satisfaction assessed by an ordinal questionnaire designed based on the Treatment Satisfaction Questionnaire for Medication (TSQM). | 42 hours
  Satisfaction assessed by an ordinal questionnaire (1 to 5, as 1 the lowest satisfaction and 5 the highest satisfaction),based on the TSQM (Treatment Satisfaction Questionnaire for Medication) version 1.4 to provide data regarding the degree of satisfaction and sensation of parents and children in relation to treatment.
Rate of Compliance comparing passive occlusion vs active occlusion (with action video games) assessed by Google Analytics and written questionnaire. | Baseline and 14h, 28h and 42 hours.
  Rate of Compliance assessed through the registration of parent-reported adherence and log file data in Google Analytics (descriptive scale of time in hours/day) for active group and parent's questionnaire for passive group (subjective scale in hours/day)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Asensio Jurado, MsC, Principal Investigator — Universitat Politècnica de Catalunya; Marc Argilés Sans, PhD, Study Director — Universitat Politècnica de Catalunya; Lluïsa Quevedo i Junyent, PhD, Study Director — Universitat Politècnica de Catalunya
Locations (1):
- Laura Asensio Jurado, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bavelier D, Green CS, Pouget A, Schrater P. Brain plasticity through the life span: learning to learn and action video games. Annu Rev Neurosci. 2012;35:391-416. doi: 10.1146/annurev-neuro-060909-152832. PMID 22715883
- [Background] Li RW, Ngo C, Nguyen J, Levi DM. Video-game play induces plasticity in the visual system of adults with amblyopia. PLoS Biol. 2011 Aug;9(8):e1001135. doi: 10.1371/journal.pbio.1001135. Epub 2011 Aug 30. PMID 21912514
- [Background] Bediou B, Adams DM, Mayer RE, Tipton E, Green CS, Bavelier D. Meta-analysis of action video game impact on perceptual, attentional, and cognitive skills. Psychol Bull. 2018 Jan;144(1):77-110. doi: 10.1037/bul0000130. Epub 2017 Nov 27. PMID 29172564
- [Background] Gambacorta C, Nahum M, Vedamurthy I, Bayliss J, Jordan J, Bavelier D, Levi DM. An action video game for the treatment of amblyopia in children: A feasibility study. Vision Res. 2018 Jul;148:1-14. doi: 10.1016/j.visres.2018.04.005. Epub 2018 May 12. PMID 29709618